CLINICAL TRIAL: NCT03360331
Title: Effect of Phosphorus on Valvular and Vascular Calcification in ESRD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Gamal Abdelmalik, Doctor, Assiut University
Other Study IDs: calcification in ESRD
Record Dates: First submitted 2017-11-05; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-10

CONDITIONS: Vascular Calcification
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the calcifying effect of phosphorus on vascular smooth muscle and detect the association between serum phosphorus and valvular and vascular calcification in end stage renal disease patients

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the main cause of death in patients with end stage renal disease(ESRD). It is estimated that ESRD patients are 5 to 20 times more likely to die because of cardiovascular causes than the general population .

Traditional cardiovascular risk factors do not completely explain higher mortality rates among hemodialysis patients , and non traditional risk factors such as anemia, bone mineral disease, hyperhomocysteinemia, inflammation, hypercoagulability, and left ventricular hypertrophy (LVH) have been demonstrated to play an important role in this population.

A number of factors have been associated with progression of vascular calcification(VC) in dialysis patients. Associations with age and duration of dialysis , diabetes mellitus ,abnormalities of mineral metabolism as well as use and dose of calcium based phosphate binders have all been reported.

Hyperphosphatemia is a common problem among patients with ESRD. It is a highly prevalent condition, as almost 40% of the U.S. hemodialysis population has a serum phosphate( PO4) greater than 6.5 mg/dl . The overall mortality risk associated with serum phosphate( PO4) above 6.5 mg/dl was 27% greater than that of patients with PO4 levels between 2.4 and 6.5 mg/dl. It is speculated that elevate PO4 may aggravate the effects of coronary atherosclerosis through increased vascular calcification and smooth muscle proliferation . It has also been suggested that myocardial calcification, a consequence of elevated PO4, may alter microcirculatory hemodynamics through increased extravascular resistance and further compromise myocardial perfusion. We, therefore, hypothesized that the increased mortality risk associated with elevated PO4 levels was primarily related to cardiac rather than non-cardiac causes of death.

A number of non-invasive imaging techniques are now available to detect and quantify vascular calcification (VC). Indeed, plain x-rays of abdomen and extremities to identify macroscopic calcifications of aorta and peripheral arteries;echocardiography for assessment of valvular calcification;2D-ultrasound for calcification of carotid arteries, femoral arteries and aorta and computed tomography technologies constitute the current armamentarium for detection and quantification of cardiovascular calcification (VC) and its progression.

Electron beam computed tomography (EBCT) and multi-slice computed tomography (MSCT) represent the gold standard for assessing the extent of coronary artery and aorta calcification.MSCT is more widely available than EBCT

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients on regular dialysis of five years duration aging 18 to 40 years

Exclusion Criteria:

* patients with hypercalcemia or hyperlipidemia or diabetic patients

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: ESRD patients on regular dialysis for five years duration aging 18 to40 years old
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Decrease the cardiovascular complications in ESRD patients | one year
  Find the relationship between phosphorus and valvular and vascular calcification in ESRD PATIENTS